CLINICAL TRIAL: NCT00145548
Title: Pilot Study of the Spiration IBV™ System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR-0003
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2007-05

CONDITIONS: Emphysema
Keywords: COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Intra Bronchial Valve

SUMMARY:
The Spiration Intra-Bronchial Valve is intended for use as a minimally invasive treatment for severe emphysema, using standard bronchoscopy. The valve is designed to limit airflow to a selected portion of the lung, producing a reduction in lung volume, which may improve pulmonary function in patients with emphysema.

DETAILED DESCRIPTION:
This pilot study is an open enrollment, prospective study with each subject serving as their own control. The sponsor may attempt to include the data from this study in the statistical analysis of the pivotal study. This proposal shall be evaluated at the conclusion of the pilot study.

PATIENT POPULATION Patients with severe emphysema are eligible to be screened for enrollment in this study. In this initial pilot study, eligible subjects will have severe, heterogeneous, predominantly upper lobe emphysema, as defined by the American Thoracic Society (ATS) 1 and the NETT Research Group.2

These subjects also will be patients who have been screened as potential candidates for LVRS, but who have been excluded from surgical treatment due to a failure to satisfy the inclusion and exclusion criteria established by the NETT Research Group for LVRS.2 Patients also will be able to tolerate a flexible bronchoscopy procedure.

Patients who have been screened and accepted for a lung transplant procedure or LVRS, and are currently registered or scheduled for such a procedure, are not eligible for enrollment in this pilot study.

Patients with an FEV1 < 20% predicted and either homogeneous emphysema or DLCO < 20% will be excluded from enrollment in this pilot study.3

Patients will be screened and enrolled until up to 115 subjects have undergone treatment with the IBV System. Up to 15 clinical centers will be selected to enroll and treat subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects at least 18 years of age.
* Subject has severe, heterogeneous, predominantly upper lobe emphysema.
* Subject has ability to meet goals of, or currently satisfies goals of, a comprehensive pulmonary rehabilitation program.
* Subject has satisfied requirement for post-rehabilitation 6-minute walk of ≥ 140 m 6 and is able to complete 3 min unloaded pedaling in exercise tolerance test.
* Subject has abstained from cigarette smoking for 4 months, as confirmed by urine or serum cotinine test.
* Pulmonary function testing results demonstrate:

  * FEV1 ≤ 45% predicted (≥ 15% predicted if age ≥ 70 years)
  * TLC ≥ 100% predicted
  * RV ≥ 150% predicted
* Arterial blood gas level indicates:

  * PCO2 ≤ 50 mm Hg
  * PO2 ≥ 45 mm Hg on room air (Denver criterion: PO2 ≥ 30 mm Hg)
* Subject has no co-existing major medical problems that would significantly increase the risk of the bronchoscopy procedure and is classified as ASA Class P4 or lower.
* If female, subject is not pregnant by a negative HCG pregnancy test within 7 days prior to the procedure.
* Subject has willingness to undertake the risk and morbidity associated with the required bronchoscopic procedures.
* Subject has willingness to participate in the study and complete the required follow-up visits.
* Subject has ability to provide informed consent.
* Subject has provided consent for treatment under this protocol and has granted access to relevant medical records to the sponsor, the Principal Investigator, the institution, the IRB and the FDA pertaining to their current lung disease condition, evaluation process, and the surgical procedure.

Exclusion Criteria:

* Patients with FEV1< 20% predicted and either homogeneous emphysema or DLCO < 20%. 3
* Subject is unable to provide informed consent.
* Subject is not an appropriate candidate for, or unable to tolerate, flexible bronchoscopy procedures.
* Subject has dysrhythmia that might pose a risk during exercise or training.
* Subject has resting bradycardia (< 50 beats/min); frequent multifocal PVCs; complex ventricular arrhythmia; sustained SVT.
* Subject has history of exercise-related syncope.
* Subject has uncontrolled hypertension (systolic, > 200 mm; diastolic > 110 mm).
* Subject has history of recurrent infections with clinically significant sputum production
* Subject has known, active asthma, chronic bronchitis or clinically significant bronchiectasis.
* Subject has giant bulla (> 1/3 volume of lung).
* Subject has pulmonary hypertension: peak systolic PPA, ≥ 45 mm Hg (Denver criterion: ≥ 50 mm Hg) or mean PPA, ≥ 35 mm Hg (Denver criterion: ≥ 38 mm Hg). (Right heart catheter is required to rule out pulmonary hypertension if peak systolic PPA on echocardiogram is ≥ 45 mm Hg.)
* Subject has requirement for > 6 L O2 to keep saturation ≥ 90% with exercise.
* Subject has evidence of systemic disease or neoplasia expected to compromise survival during the 1-year study period.
* Subject demonstrates 6MWT distance ≤ 140 m after rehabilitation.
* Subject has any disease or condition that interferes with completion of initial or follow-up assessments.
* Subject has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.
* Subject has only the homogeneous emphysema pattern.
* Subject is classified as ASA Class greater than P4 7 including presence of co-morbidity that could significantly increase the risk of a standard bronchoscopy procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2003-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is to evaluate the safety of the device, during deployment and short-term implantation for a period of up to 3 months.

SECONDARY OUTCOMES:
The secondary endpoint is to estimate the effectiveness achieved after 1 and 3 months of use.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Emory Health Care, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Lahey Clinic, Burlington, Massachusetts
  - North Shore - Long Island Jewish Health System, Long Island City, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Coxson HO, Nasute Fauerbach PV, Storness-Bliss C, Muller NL, Cogswell S, Dillard DH, Finger CL, Springmeyer SC. Computed tomography assessment of lung volume changes after bronchial valve treatment. Eur Respir J. 2008 Dec;32(6):1443-50. doi: 10.1183/09031936.00056008. Epub 2008 Aug 6. PMID 18684848
- See also: Related Info — http://www.spiration.com